CLINICAL TRIAL: NCT02006069
Title: MOre REsponse on Cardiac Resynchronization Therapy (CRT) With MultiPoint Pacing (MPP)
Brief Title: MOre REsponse on Cardiac Resynchronization Therapy With MultiPoint Pacing
Acronym: MORE CRT MPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The steering committee had decided to discontinue enrollment because the interim analysis showed a low probability that the study would meet the primary endpoint. The interim analysis did not demonstrate any safety concerns with activating MPP.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-13-006-ID-HF
Record Dates: First submitted 2013-09-23; First posted 2013-12-09 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
Keywords: CRT, non responders, MultiPoint Pacing (MPP)
MeSH Terms: conditions — Heart Failure; Creatine deficiency, X-linked

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MPP ON (Experimental): MPP ON: feature is enabled
  Interventions: Device: MPP
- MPP OFF (No Intervention): MPP OFF: feature not enabled

INTERVENTIONS:
Device: MPP — All patients enrolled in the study will be implanted (according to current Guidelines) with an MPP compatible CRT device.
  The MPP feature will be evaluated in two study phases. Patients randomized to MPP in Phase I will have MPP programmed per the physician's discretion ("no mandated MPP programming") and patients randomized to MPP in Phase II will have MPP programmed per protocol requirements ("mandated MPP programming").
  Arms: MPP ON

SUMMARY:
The purpose of this Clinical investigation is to assess the impact of the Multi Point Pacing (MPP) feature at 12 months in the treatment of patients not responding to standard Cardiac Resynchronization Therapy (CRT) after 6 months.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, multi-center trial. Data will be collected at enrollment, baseline, implant procedure, patient classification, 6 months and 12 months of follow-up. During the 6-month visit, the patient's response to CRT will be evaluated according to LVESV reduction. Patients with an LVESV reduction of at least 15% will be classified as responders. These patients will terminate their participation in the study and return to the center's standard practice. Patients with an LVESV reduction less than 15% will be classified as non-responders and the MPP feature will be activated according to randomization result and they will be followed until the 12-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Meets the current ESC Guidelines or ACCF/AHA/HRS Class I or Class IIa indications for CRT implant (including upgrades from single or dual chamber ICDs)
* Must be willing and able to comply with study requirements
* Must indicate their understanding of the study and willingness to participate by signing an appropriate informed consent form

Exclusion Criteria:

* Already had a CRT device implanted
* Myocardial Infarction, unstable angina within 40 days prior the enrollment
* Recent cardiac revascularization (PTCA, Stent or CABG) in the 4 weeks prior to enrollment or planned for the 3 months following
* Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) in the 3 months prior the enrollment
* Primary valvular disease
* Atrial Fibrillation:

  * Persistent AF at the time of enrollment
  * Permanent AF not treated with AV node ablation within 2 weeks from the CRT implant
  * History or incidence of Paroxysmal or Persistent AF within 30 days prior the enrollment
* Unable to comply with the follow up schedule
* Less than 18 years of age
* Pregnant or are planning to become pregnant during the duration of the investigation
* Classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 12 months
* Undergone a cardiac transplantation
* Life expectancy < 12 months
* Currently participating in any other clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5850 (Actual)
Dates: Start 2013-12; Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Leclercq, Study Chair — Centre Cardio-Pneumologique, CHU Pontchaillou
Locations (206):
- United States (32):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Comprehensive Cardiovascular, Bakersfield, California
  - Glendale Adventist Medical Center, Glendale, California
  - Scripps Health, La Jolla, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Cardiac Rhythm Specialists, Inc., Reseda, California
  - San Diego Cardiac Center, San Diego, California
  - Colorado Heart & Vascular, P.C., Lakewood, Colorado
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Coliseum Medical Centers, Macon, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - St. Elizabeth Medical Center - South Unit, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - McLaren Health Care Corporation, Auburn Hills, Michigan
  - MidMichigan Medical Center-Midland, Midland, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - CHI Health Creighton University Medical Center-Bergan Mercy, Omaha, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Cardiology Associates of Fairfield County, PC, Haddon Heights, New Jersey
  - Samaritan Heart & Vascular Institute - Cardiology Dept., Corvallis, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Francis Hospital, Greenville, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Memorial Katy Cardiology Associates, Houston, Texas
  - Vivek Mangla, MD, Lufkin, Texas
  - EP Heart, The Woodlands, Texas
- Australia (5):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Bedford Park
  - St. Andrews War Memorial Hospital, Brisbane
  - The Alfred Hospital, Melbourne
  - Westmead Hospital, Westmead
- Austria (3):
  - Krankenhaus der Stadt St. Poelten, Sankt Pölten
  - Krankenhaus Hietzing, Vienna
  - Wilhelminenspital, Vienna
- Belgium (2):
  - Hopital Erasme, Brussels
  - St. Joseph Gilly, Gilly
- Canada (12):
  - Foothills Medical Centre, Calgary
  - Royal Alexandra Hospital, Edmonton
  - QEII Health Sciences, Halifax
  - Kingston General Hospital, Kingston
  - Hôtel Dieu de CHUM, Montreal
  - Institut de Cardiologie de Montreal, Montreal
  - McGill University Health Centre General Hospital, Montreal
  - Institut de Cardiologie de Quebec, Sainte-Foy
  - CHUS Fleurimont, Sherbrooke
  - HSC, Eastern Health, St. Johns
  - Rouge Valley Centenary, Toronto
  - St. Paul's Hospital, Vancouver
- Prince of Wales Hospital, Hong Kong, China
- Colombia (2):
  - Angiografia Clinica de Occidente, Cali
  - Clínica Cardio VID, Medellín
- Denmark (3):
  - Odense University Hospital, Odense, Fyn
  - Aalborg Sygehus Syd, Aalborg, North Denmark
  - Skejby University Hospital, Aarhus
- Finland (2):
  - Keski-Suomi Central Hospital, Jyväskylä
  - Turku University Hospital, Turku
- France (21):
  - Hôpital Clairval, Marseille, Alpes
  - CHU Cavale Blanche, Brest
  - CHU Trousseau, Chambray-lès-Tours
  - CHU François Mitterrand Dijon Bourgogne, Dijon
  - CHRU Albert Michallon, Grenoble
  - CHRU Lille, Lille
  - Hopital Saint Philibert, Lomme
  - Hôpital Saint Joseph, Marseille
  - Centre Hospitalier de Belfort-Montbeliard, Montbéliard
  - CHU Montpellier, Montpellier
  - CHU de Nancy - Hopital de Brabois, Nancy
  - CHU Hopital G. & R. Laënnec, Nantes
  - Nouvelles cliniques Nantaises, Nantes
  - Centre Cardiologique Du Nord, Paris
  - Hopital Pitiè Salpetrière, Paris
  - Institute Cardio. Paris-Sud - Institut Jacques Cartier, Paris
  - CHRU Hôpital de Pontchaillou, Rennes
  - CHRU Rouen Hospital Charles Nicolle, Rouen
  - CHR de La Reunion - Site du CHFG, Saint-Denis
  - Centre Hospitalier de Valence, Valence
  - Clinique du Tonkin, Villeurbanne
- Germany (33):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Hegau-Bodensee-Hochrhein-Kliniken GmbH, Singen, Baden-Wurttemberg
  - Kerckhoff-Klinik gGmbH, Bad Nauheim, Hesse
  - Herz- und Gefäßzentrum am Krankenhaus Neu-Bethlehem, Göttingen, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Medizinische Einrichtungen der Universität zu Köln, Cologne, North Rhine-Westphalia
  - Evangelisches Krankenhaus Kalk gGmbH, Cologne, North Rhine-Westphalia
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
  - Schuchtermann-Schillersche Kliniken, Bad Rothenfelde
  - Charite Campus Virchow Klinikum, Berlin
  - Universitatsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - Klinikum Bielefeld, Bielefeld
  - Berufsgenossenschaftliche Kliniken Bergmannsheil, Bochum
  - Klinikum Coburg, Coburg
  - St. Vinzenz-Hospital, Cologne
  - Helios-Klinikum Erfurt GmbH, Erfurt
  - Kliniken der Friedrich-Alexander-Universität, Erlangen
  - Elisabeth-Krankenhaus Essen GmbH, Essen
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Universitatsklinikum Greifswald, Greifswald
  - Klinikum Gütersloh gGmbH, Gütersloh
  - Albertinen-Krankenhaus Hamburg, Hamburg
  - Klinikum Ingolstadt, Ingolstadt
  - Klinikum St. Georg gGMbH, Leipzig
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum Ludenscheid, Lüdenscheid
  - St.-Marien-Hospital GmbH, Lünen
  - Deutsches Herzzentrum München des Freistaates Bayern, München
  - Universitatsklinikum Muenster, Münster
  - Klinikum Oldenburg, Oldenburg
  - Krankenhaus der Barmherzigen Bruder, Trier
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen
  - Universitätsklinikum Würzburg, Würzburg
- The Onassis Cardiac Center, Athens, Greece
- India (8):
  - Medanta - The Medicity Hospital, Gurgaon, Haryana
  - Fortis Hospital, Bangalore, Karnataka
  - Care Institute of Medical Sciences, Ahmedabad
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Apollo Hospital, Chennai
  - CARE Banjara, Hyderabad
  - Medanta Medicity Hospital, New Delhi
  - Escorts Heart Institute and Research Centre, New Delhi
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Medical Center, Tel Aviv
- Italy (21):
  - Az.Osp.Universitaria Consorziale Policlinico, Bari
  - Azienda Ospedaliera Di Venere, Bari
  - Policlinico S.Orsola Malpighi, Bologna
  - Az. Osp. Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera S. Anna e S Sebastiano, Caserta
  - Presidio Osp. Vito Fazzi, Lecce
  - Clinica Mediterranea, Naples
  - Ospedale dei Pellegrini, Naples
  - Ospedale S. Giovanni Bosco, Naples
  - Az Osp.Universitaria Maggiore della Carità, Novara
  - Università degli Studi di Padova, Padua
  - Casa di Cura Dott. Pederzoli, Peschiera del Garda
  - Az. Osp. Universitaria Pisana-Presidio Santa Chiara, Pisa
  - Ospedale di Portogruaro, Portogruaro
  - Azienda Ospedaliera "Civile - Maria Paternò Arezzo", Ragusa
  - Ospedale Madre G. Vannini, Roma
  - Policlinico Casilino, Roma
  - Ospedale S. Giovanni Calibita Fatebenefratelli di Roma, Rome
  - Azienda Ospedaliera S. Anna, San Fermo della Battaglia
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale Civile Maggiore di Verona Borgo Trento, Verona
- American University of Beirut Medical Center, Beirut, Lebanon
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Mater Dei Hospital, Paola, Malta
- Netherlands (5):
  - Twee Steden Ziekenhuis, Tilburg, North Brabant
  - Amsterdam Academic Medical Center (AMC), Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Isala Ziekenhuis, Zwolle
- Poland (4):
  - Szpital Kliniczny Premienienia Panskiego, Poznan, Greater Poland Voivodeship
  - Gornoslaskie Centrum Medyczne im.prof. Leszka Gieca, Katowice, Silesian Voivodeship
  - Slaskie Centrum Chorob Serca, Zabrze, Silesian Voivodeship
  - Wojewodzki Specjalistyczny Szpital im. Bieganskiego, Lodz
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar do Alto Ave, Unidade de Guimarães, Creixomil
  - Hospital de Santa Cruz, Lisbon
  - Hospital Garcia de Orta, EPE, Lisbon
  - Santa Maria Hospital, Lisbon
  - Centro Hospitalar Vila Nova Gaia, Vila Nova de Gaia
- Puerto Rico (2):
  - Arrhythmia Group, Ponce
  - Heart Rhythm Management, San Juan
- Saudi Arabia (2):
  - King Fahad Armed Forces Hospital, Jeddah
  - King Fahad Medical City, Riyadh
- National University Hospital, Singapore, Singapore
- South Korea (6):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul St. Mary's Hospital, Seoul, Seocho-gu
  - Sejong General Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
- Spain (14):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital de la Santa Creu y Sant Pau, Barcelona
  - Hospital Universitario Virgen de la Nieves, Granada
  - Complexo Hospitalario Universitario de Santiago, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - HCU Virgen de la Victoria, Málaga
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Alvaro Cunqueiro, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- Karolinska University Hospital Huddinge, Stockholm, Sweden
- Hopital Cantonal Universitaire de Geneva, Geneva, Switzerland
- Taiwan (2):
  - National Taiwan University, Taipei City, Taipei
  - Chang Gung Memorial Hospital, Linkou District
- United Kingdom (10):
  - Wansbeck General Hospital, Ashington
  - Queen Elizabeth Hospital, Birmingham
  - The Royal Sussex Country Hospital, Brighton
  - Golden Jubilee National Hospital, Glasgow
  - Kings College Hospital, London
  - St. Thomas Hospital, London
  - Manchester Heart Center, Manchester Royal Infirmary, Manchester
  - John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southampton
  - The Great Western Hospital, Swindon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leclercq C, Burri H, Curnis A, Delnoy PP, Rinaldi CA, Sperzel J, Lee K, Calo L, Vicentini A, Concha JF, Thibault B. Cardiac resynchronization therapy non-responder to responder conversion rate in the more response to cardiac resynchronization therapy with MultiPoint Pacing (MORE-CRT MPP) study: results from Phase I. Eur Heart J. 2019 Sep 14;40(35):2979-2987. doi: 10.1093/eurheartj/ehz109. PMID 30859220
- [Derived] Leclercq C, Burri H, Curnis A, Delnoy PP, Rinaldi CA, Sperzel J, Lee K, Cohorn C, Thibault B; MORE-CRT MPP Investigators. Rationale and design of a randomized clinical trial to assess the safety and efficacy of multipoint pacing therapy: MOre REsponse on Cardiac Resynchronization Therapy with MultiPoint Pacing (MORE-CRT MPP-PHASE II). Am Heart J. 2019 Mar;209:1-8. doi: 10.1016/j.ahj.2018.12.004. Epub 2018 Dec 8. PMID 30616009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled eligible patients with a standard CRT indication after obtaining written informed consent. The implanting physician programmed biventricular pacing (BiVP) at implant in those patients who had the quadripolar CRT system successfully implanted The implanting physician programmed the LV pacing vector, A-V delay, and V-V delay settings at their discretion until the patient's randomization at 6 months.
Pre-assignment Details: For the first 6 months post-implant, all enrolled patients were followed with traditional biventricular pacing (BiVP). Only patients not responding to BiVP between baseline and 6 months (using LVESV reduction less than 15%), which is called CRT non-responders, were randomized to either MPP or continuous BiVP arm at 6 months and followed until 12 months.
Groups:
- MPP ON: MPP ON: feature is enabled after 6 months
  MPP: All patients enrolled in the study will be implanted (according to current Guidelines) with an MPP compatible CRT device.
  The MPP feature will be evaluated in two study phases. Patients randomized to MPP in Phase I will have MPP programmed per the physician's discretion ("no mandated MPP programming") and patients randomized to MPP in Phase II will have MPP programmed per protocol requirements ("mandated MPP programming").
- BiVP: MPP OFF: Continuous BiVP after 6 months
Period: Overall Study
Arm/Group | MPP ON | BiVP
Started | 510 | 558
Completed | 271 | 555
Not Completed | 239 | 3
Not completed — MPP other programming | 239 | 0
Not completed — RV only pacing | 0 | 3

BASELINE CHARACTERISTICS:
Population: A race/ethnicity baseline was not collected in the study.
Groups:
- MPP ON: MPP ON: feature is enabled after 6 months
  MPP: All patients enrolled in the study will be implanted (according to current Guidelines) with an MPP compatible CRT device. The MPP feature was evaluated in two study phases. Patients randomized to MPP in Phase I had MPP programmed per the physician's discretion ("no mandated MPP programming") and patients randomized to MPP in Phase II had MPP programmed per protocol requirements ("mandated MPP programming"). Patients from both Phases were analyzed together using as-treated analysis.
- BiVP: MPP OFF: Continuous BiVP after 6 months. Patients from both Phases were analyzed together using as-treated analysis.
- Total: Total of all reporting groups
Arm/Group | MPP ON | BiVP | Total
Number analyzed (Participants) | 271 | 555 | 826
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.3) | 68.1 (10.6) | 68.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 123 | 168
  Male | 226 | 432 | 658
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Cardiomyopathy [Count of Participants; unit: Participants]
  Ischemic | 147 | 278 | 425
  Non-ischemic | 124 | 277 | 401
NYHA Class [Count of Participants; unit: Participants] — Class I: No limitation of physical activity Class II(Mild): Slight limitation of physical activity. Class III(Moderate): Marked limitation of physical activity. Class IV(Severe): Unable to carry out any physical activity without discomfort.
  Increasing functional class is associated with greater risk of death and hospitalization.
  Participants
    II | 129 | 272 | 401
    III | 137 | 268 | 405
    IV | 4 | 13 | 17
    Not done | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Non-responder Patients Who Converted to Responders
Description: The primary endpoint of this study is evaluated at 12 months after enrollment and it is defined as the percentage of non-responder patients converted to responders after 6 months of MPP feature turned ON compared to baseline, as measured by Left Ventricular End Systolic Volume (LVESV) reduction of at least 15%.
Time Frame: Non-responder to responder conversion rate between randomization at 6 months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MPP ON | BiVP
Number analyzed (Participants) | 271 | 555
Participants | 84 | 170

2. Secondary Outcome: Reduction of Left Ventricular End-systolic Volume (LVESV) in Acute Phase
Description: Reduction of LVESV between baseline and 6 Months visit
Time Frame: Baseline vs 6 Months
Measure: Mean (Standard Deviation); unit: percentage of LVESV change
Arm/Group | MPP ON | BiVP
Number analyzed (Participants) | 271 | 555
percentage of LVESV change | 2.1 (11.2) | 0.1 (3.3)

3. Secondary Outcome: Clinical Composite Score Evaluation
Description: Packer's Clinical Composite Score evaluation between baseline and 12 months as defined below,
  * Worsened: the patient died because of cardiovascular reasons OR experienced a HF event OR demonstrated worsening in NYHA functional class, or had worsening of patient global assessment (PGA) score compared with the last observation
  * Improved: the patient survived without an HF event AND demonstrated either improvement in NYHA functional class or improvement in PGA score or both compared with the last observation
  * Unchanged: the patient was neither improved nor worsened
Time Frame: Baseline vs 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MPP ON | BiVP
Number analyzed (Participants) | 271 | 555
Participants
  Improved | 161 | 312
  Unchanged | 56 | 124
  Worsensed | 54 | 119

4. Secondary Outcome: Reverse Left Ventricular (LV) Remodeling
Description: Evaluation of Reverse LV remodeling, measured as changed in left ventricular end-systolic volume (LVESV) from baseline to 12 months
Time Frame: Baseline vs 12 Months
Population: Only subjects with LVESV data available at both baseline and 12 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MPP ON | BiVP
Number analyzed (Participants) | 267 | 538
mL | 3.0 (24) | 3.8 (23.1)

5. Secondary Outcome: NYHA Class Changes
Description: Evaluation of NYHA Class changes between baseline and 12 months. Increasing functional class is associated with greater risk of death or hospitalization.
Time Frame: Baseline vs 12 Months
Population: Only subjects with NYHA data available at both baseline and 12 months were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MPP ON | BiVP
Number analyzed (Participants) | 266 | 532
Participants
  Improved | 125 | 287
  Unchanged | 129 | 225
  Worsened | 12 | 20

6. Secondary Outcome: 6MWT Changes
Description: Evaluation of the patient's activity status using 6 Minutes Walking Test changes from baseline to 12 months FU
Time Frame: Baseline vs 12 Months
Population: Only subjects with 6MHWT data available at both baseline and 12 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MPP ON | BiVP
Number analyzed (Participants) | 221 | 441
meters | 41.1 (113.6) | 46 (121.1)

7. Secondary Outcome: Patient's QoL Score Changes (MLWHF)
Description: Evaluation of patient's Quality of Life score using Minnesota Living with Heart Failure (MLWHF) Questionnaires. The MLWHF Questionnaire consists of 21 questions with a range in overall scores of 0 to 105 points (lower scores indicate better quality of life).
Time Frame: Baseline vs 12 Months
Population: Only subjects with MLWHF data available at both baseline and 12 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MPP ON | BiVP
Number analyzed (Participants) | 261 | 523
score on a scale | -11.6 (20.0) | -12.2 (21.7)

ADVERSE EVENTS:
Time Frame: 6 months to 12 months after randomization
Arm/Group | MPP ON | BIVP
All-Cause Mortality (participants affected / at risk) | 4/271 | 18/555
Serious Adverse Events (participants affected / at risk) | 82/271 | 190/555
Other Adverse Events (participants affected / at risk) | 67/271 | 118/555
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPP ON (N=271) | BIVP (N=555)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anticoagulant Overdose (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Atrial or Ventricular Arrhythmia (Cardiac disorders) | 23 (28) | 42 (60)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 3 (4)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorespiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 5 (5)
Dyspnea (Cardiac disorders) | 0 (0) | 2 (2)
Exacerbation of Heart Failure (Cardiac disorders) | 30 (40) | 53 (76)
Heart Block (Cardiac disorders) | 0 (0) | 1 (1)
Mitral Valve Dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 2 (4) | 3 (3)
Pacemaker Mediated Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pain (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (2)
Pulmonary Edema (Cardiac disorders) | 4 (5) | 7 (8)
Sudden Cardiac Death (Cardiac disorders) | 0 (0) | 1 (1)
Valve Damage (Cardiac disorders) | 1 (1) | 3 (3)
Exacerbation of Heart Failure (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism Caused by Amiodarone (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal Affliction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding/Hematoma/Seroma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Downhill Varicose and Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal Varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal Disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Obstipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic Cystic Lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug Side Effect (General disorders) | 1 (1) | 0 (0)
Infection (General disorders) | 0 (0) | 1 (1)
Nausea, Vomiting (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Pain at Pulse Generator Site (General disorders) | 1 (1) | 0 (0)
Gallbladder Disease (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug Allergy (Immune system disorders) | 0 (0) | 1 (1)
Interstitial Pulmonary Fibrosis (Immune system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 7 (8) | 16 (21)
Bleeding/Hematoma/Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bone Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac Perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Infection (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Mild Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain at Pulse Generator Site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pericardial Effusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Pocket Swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Subdural Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte Disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid Accumulation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myogelosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6)
Ureteral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellar Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 3 (3) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal Lead Pacing Impedance <= 200 OHMS or >=2000 OHMS (Product Issues) | 1 (1) | 0 (0)
Elevated Pacing Thresholds/Loss of Capture (Product Issues) | 0 (0) | 1 (1)
Extracardiac Stimulation (Phrenic Nerve, Diaphragm, Chest Wall) (Product Issues) | 1 (1) | 1 (1)
Infection (Product Issues) | 1 (1) | 0 (0)
Lead Dislodgement or Migration (Product Issues) | 8 (9) | 36 (40)
Lead Fracture (Product Issues) | 0 (0) | 1 (1)
Oversensing (Product Issues) | 0 (0) | 2 (2)
Pulse Generator Migration (Product Issues) | 0 (0) | 1 (1)
Therapy for Non-Ventricular Rhythm (Product Issues) | 1 (1) | 2 (4)
Undersensing (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Dementia (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep Apnea (Psychiatric disorders) | 0 (0) | 3 (4)
Kidney Disease (Renal and urinary disorders) | 4 (4) | 11 (12)
Renal Disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary Tract Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Larynx Perforation After Tee (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pseudo-Nodular Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Limb Gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bone Fracture (Surgical and medical procedures) | 0 (0) | 1 (1)
Nose Resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Bleeding/Hematoma/Seroma (Vascular disorders) | 6 (7) | 9 (9)
Bypass Graft Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Intracardiac Thrombus (Vascular disorders) | 0 (0) | 1 (1)
Lower Extremity Claudication (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Artery Disease (Vascular disorders) | 1 (1) | 2 (2)
Syncope (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
TIA (Vascular disorders) | 0 (0) | 1 (1)
Venous Occlusion (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPP ON (N=271) | BIVP (N=555)
Atrial or Ventricular Arrhythmia (Cardiac disorders) | 24 (29) | 41 (43)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
Exacerbation of Heart Failure (Cardiac disorders) | 5 (7) | 13 (13)
Heart Transplant (Cardiac disorders) | 0 (0) | 1 (1)
Pacemaker Mediated Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyreosis (Endocrine disorders) | 1 (1) | 0 (0)
Chest Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mild Diverticulosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pain at Pulse Generator Site (General disorders) | 1 (1) | 2 (2)
Worsening of General Patient's Condition (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 4 (4)
Bone Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Bodily Rejection Phenomena (Product Issues) | 0 (0) | 1 (1)
Elevated Pacing Thresholds/Loss of Capture (Product Issues) | 5 (6) | 8 (9)
Extracardiac Stimulation (Phrenic Nerve, Diaphragm, Chest Wall) (Product Issues) | 13 (16) | 26 (31)
Lead Dislodgement or Migration (Product Issues) | 3 (3) | 2 (2)
Oversensing (Product Issues) | 3 (3) | 5 (6)
Pacemaker Mediated Tachycardia (Product Issues) | 1 (1) | 0 (0)
Palpitation (Product Issues) | 1 (1) | 0 (0)
Therapy for Non-Ventricular Rhythm (Product Issues) | 2 (2) | 2 (2)
Sleep Apnea (Psychiatric disorders) | 1 (1) | 0 (0)
Kidney Disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elective Replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Bleeding/Hematoma/Seroma (Vascular disorders) | 1 (1) | 10 (10)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)
Syncope (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous Occlusion (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT02006069/Prot_SAP_000.pdf